CLINICAL TRIAL: NCT01199770
Title: Understanding Pasta Formulations and Portion Size on Satiety in Healthy Weight Women
Brief Title: Pasta Formulations, Portion Sizes and Their Effect on Appetite
Acronym: SET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: Barilla America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SET 2010-043
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Healthy; Appetite
Keywords: pasta; appetite; hunger; satiety; nutrition; metabolic; gut peptide hormones; psychological phenomena and processes
MeSH Terms: interventions — Culture Media

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- experimental pasta B, small (Experimental): small portion experimental pasta B
  Interventions: Other: Experimental B, small
- experimental pasta C, small portion (Experimental): small portion experimental pasta C
  Interventions: Other: Experimental pasta C, small
- Control pasta, small (Placebo Comparator): small portion Control pasta
  Interventions: Other: Control, small
- No Load (Other): Only water
  Interventions: Other: NL
- Control pasta, medium (Active Comparator): medium portion Control pasta
  Interventions: Other: control, medium
- experimental pasta B, medium portion (Experimental): medium portion experimental pasta B
  Interventions: Other: experimental pasta B, medium
- experimental pasta C, medium portion (Experimental): medium portion experimental pasta B
  Interventions: Other: experimental pasta C, medium

INTERVENTIONS:
Other: Control, small — control pasta, small portion
  Arms: Control pasta, small
Other: Experimental B, small — experimental pasta, small portion
  Arms: experimental pasta B, small
Other: Experimental pasta C, small — experimental pasta C, small portion
  Arms: experimental pasta C, small portion
Other: control, medium — control pasta, medium portion
  Arms: Control pasta, medium
Other: experimental pasta B, medium — experimental pasta B, medium portion
  Arms: experimental pasta B, medium portion
Other: experimental pasta C, medium — experimental pasta C, medium portion
  Arms: experimental pasta C, medium portion
Other: NL — no pasta, water only
  Arms: No Load

SUMMARY:
Investigators are interested in learning how appetite responds to pasta containing different amounts of protein and fiber when provided in two different portion sizes.

In this research study, subjects will be asked to eat an entire pasta serving containing different amounts of protein and fiber mixtures. Subjects will be asked to do this on six separate occasions. One time subjects will not receive pasta, only water.

After the pasta serving, there will be a buffet of deli style lunch items and subjects may eat as much they desire. Thereafter subjects will describe their feelings of hunger, fullness and desire to eat for 3 hours. In addition, blood will be taken throughout the study period to determine how eating pasta servings in different portion sizes impacts certain hormones released from the intestine, and therefore how they influence appetite. All study visits will take approximately 4 ½ - 5 hours.

DETAILED DESCRIPTION:
The study is a randomized, 7-arm, treatment-controlled, within-subjects, 3-hour postprandial crossover study to evaluate the satiety and metabolic effects of pasta formulations in 2 portion sizes on lunch intake in healthy weight women. The study design will test 3 varying pasta formulations (2 experimental and 1 standard control) at 2 fixed portion sizes in a preload plus test lunch setting in relatively healthy unrestrained women.

This study will require one initial screening visit (approximately 1 hour) and seven study visits each lasting approximately 5 hours. All visits should be completed within 2 months. We are looking for healthy, non-smoking women older than 18 years of age with no significant medical history.

The initial screening visit will determine subject eligibility through height, weight and waist circumference measurements, vital signs, blood glucose test (finger prick) and completion of a series of surveys relating to eating, health, exercise and mood.

If willing and eligible to participate, subjects will have seven study visits. The pasta meal will be provided 5 hours after a standardized breakfast which is considered the usual breakfast for each subject at the same time of day on each study visit day. Upon arrival at each visit, subjects will have anthropometric measurements, vital signs and blood glucose finger prick. Thereafter, subjects will document subjective feelings of satiety followed by a blood draw. Upon completion of pre-study procedures, subjects will be asked to consume an entire pasta serving (with the exception of one visit, where no pasta will be served). Shortly thereafter, subjects will be served a buffet lunch and they may eat as desired, asking for more if desired. Throughout the study and after the lunch buffet, subjects will be followed for 3 hours assessing subjective feelings of satiety at designated time points along with blood draws measuring metabolic associated meal responses. During the course of the study, subjects will be instructed to maintain their usual level of activity and diet. Four day food records will be maintained throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Females
* 18 years of age and older
* Body mass index (BMI) between 18.5 and 24.9 kg/m2, inclusive
* No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Unrestrained eater (score < 10 on the Three Factor Eating Questionnaire)

Exclusion Criteria:

* Pregnant and/or lactating or planning for pregnancy
* Allergies or intolerances to foods consumed in the study
* Fasting blood glucose > 110 mg/dL. Subjects identified with elevated fasting blood glucose levels will be will be advised to contact their primary care physician for appropriate follow-up care.
* Taking over the counter fiber supplements or other supplements that may interfere with the study procedures or endpoints
* Taking prescription medications that may interfere with study procedures or endpoints ( medications that affect appetite)
* Subjects with unusual dietary habits (e.g. pica)
* Actively losing weight or trying to lose weight (unstable body weight fluctuations of > 5 kg in a 60 day period)
* Excessive exercisers or trained athletes
* Addicted to drugs and/or alcohol
* Medically documented psychiatric or neurological disturbances
* Smoker (past smoker may be allowed if cessation is > 2 years)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological sex of eligible participants
Enrollment: 24 (Actual)
Dates: Start 2010-09-15 (Actual); Primary Completion 2011-11-18 (Actual); Study Completion 2011-11-18 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of pasta formulations and portion size incorporated into a lunch meal on satiety (inhibition of further eating) as determined by subsequent second meal intake along with subjective responses on visual analog scales | 3 hour post prandial study
  Meals will be provided 4 1/2 hours after a standardized breakfast and subjects must eat the entire pasta serving. After the pasta serving, a buffet lunch will be served and subjects may eat as much as desired. Immediately thereafter, subjects will record satiety responses at 0 min (immediately post consumption), 20, 40, 60, 90, 120, 150 and 180 on a visual analog scale (VAS). The subject will answer a series of questions on the VAS at each respective time point describing their feelings of hunger, fullness and desire to eat.

SECONDARY OUTCOMES:
To investigate the effect of pasta formulations and portion size incorporated into a lunch meal on postprandial intestinal phase mechanisms of satiety and meal-associated metabolic response patterns | 3 hour postprandial study
  Meals will be provided 4 1/2 hours after a standardized breakfast and subjects must eat the entire pasta serving. After the pasta serving, a buffet lunch will be served and subjects may eat as much as desired. Immediately thereafter, subjects will have blood drawn at 0 min (immediately post consumption), 20, 40, 60, 90, 120, 150 and 180. Blood samples will be drawn for measurement of plasma lipids, glucose, insulin and gut peptide hormones (GLP-1 and PYY).

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, PhD, MS, Principal Investigator — Clinical Nutrition Research Center, Illinois Institute of Technology; Indika Edirisinghe, PhD, Principal Investigator — Clinical Nutrition Research Center, Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States